CLINICAL TRIAL: NCT01194271
Title: A Neoadjuvant Phase IIa Study of Ipilimumab {Formerly Known as MDX-010 (BMS-734016)} Plus Hormone Ablation in Men With Prostate Cancer Followed by Radical Prostatectomy.
Brief Title: Neoadjuvant Ipilimumab in Prostate Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2009-0135; NCI-2010-01974 (Registry Identifier: NCI CTRP)
Record Dates: First submitted 2010-09-01; First posted 2010-09-02 (Estimated); Results first posted 2020-09-03 (Actual); Last update posted 2024-06-06 (Actual); Status verified 2023-09

CONDITIONS: Prostate Cancer
Keywords: Hormone Ablation; Prostate adenocarcinoma; Radical prostatectomy; Leuprolide Acetate; Lupron Depot; Ipilimumab; BMS-734016; MDX010
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Leuprolide; Ipilimumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Neoadjuvant Ipilimumab (Experimental): Leuprolide Acetate 22.5 mg administered as a single intramuscular 3 month depot + Ipilimumab 10 mg/kg by vein administered as 2 single doses, 3 weeks apart after hormone therapy + Radical Prostatectomy Surgery to remove prostate gland approximately 4 weeks after the second dose of Ipilimumab.
  Interventions: Drug: Leuprolide Acetate; Drug: Ipilimumab; Procedure: Radical Prostatectomy

INTERVENTIONS:
Drug: Leuprolide Acetate — 22.5 mg administered as a single intramuscular 3 month depot.
  Other Names: Lupron Depot
Drug: Ipilimumab — 10 mg/kg by vein administered as 2 single doses, 3 weeks apart after hormone therapy.
  Other Names: BMS-734016; MDX010
Procedure: Radical Prostatectomy — Surgery to remove prostate gland approximately 4 weeks after the second dose of Ipilimumab.

SUMMARY:
The goal of this clinical research study is to learn how ipilimumab in combination with Lupron (leuprolide acetate) affects the body's own defense (immune) system before having surgery to remove prostate cancer. The safety of the drug combination will also be studied.

DETAILED DESCRIPTION:
The Study Drugs:

Ipilimumab is designed to cause an immune response in your body by blocking 2 specific molecules that usually block an immune response. This may help to kill cancer cells.

Leuprolide acetate is designed to lower the level of testosterone (a male hormone) in the blood. This may slow the growth of cancer cells.

Study Drug Administration:

If you are found to be eligible to take part in this study, you will receive a leuprolide acetate injection in your muscle. This is considered Week 0. One week later, you will begin treatment with ipilimumab. Ipilimumab will be given by vein over 90 minutes during Weeks 1 and 4 (about 21 days apart). During the infusion, your blood pressure will be measured every 30 minutes, and again an hour after you are finished receiving the drug.

Study Visits:

At Weeks 0, 1, 4 and 7, the following tests and procedures will be performed:

* You will have a physical exam, including measurement of your vital signs and weight.
* You will be asked about any drugs or treatments you may be receiving.
* You will be asked about any side effects you may have experienced.
* Your performance status will be recorded.
* Blood (about 7-10 tablespoons) will be drawn for routine tests. This blood will also be tested to measure your protein, PSA and testosterone levels, to check the function of your thyroid and adrenal glands, and to test for an immune response.

Surgery:

About 4 weeks after your second treatment with ipilimumab, you will have surgery to remove your prostate gland. You will be asked to sign a separate consent form that describes the surgery and its risks. A sample of the leftover prostate gland tissue from surgery will be tested for an immune response. On that day, the following tests and procedures will be performed:

Between 14 and 24 weeks after your surgery, you will return to the clinic for your post-operative follow-up visit. The following tests and procedures will be performed:

* You will have a physical exam, including measurement of your vital signs and weight.
* Your performance status will be recorded.
* You will be asked about any drugs or treatments you may be receiving.
* You will be asked about any side effects you have experienced since your last visit.
* Blood (about 7-10 tablespoons) will be drawn for routine tests. This blood will also be used to measure your protein, testosterone and PSA levels, to check the function of your thyroid and adrenal glands, and to test for an immune response.
* You will have a bone scan, and either a CT or MRI scan of your chest, abdomen, and pelvis to check the status of the disease.

Length of Study:

You will only receive 2 treatments with ipilimumab on this study. You will be on study until 24 weeks after surgery. You will be taken off study if intolerable side effects occur, if the disease gets worse, or if the study doctor thinks it is in your best interest to be taken off study.

This is an investigational study. Ipilimumab is not FDA approved or commercially available. Ipilimumab is currently being used for research purposes only. Leuprolide acetate is FDA approved for management of metastatic prostate cancer but is not approved for use before definitive surgery. It is commercially available to treat prostate cancer.

Up to 20 patients will take part in this study. All will be enrolled at MD Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. Willing and able to give written informed consent;
2. Histologic Documentation: Histologic documentation of prostatic adenocarcinoma. Patients with small cell, neuroendocrine, or transitional cell carcinomas are not eligible. All eligible patients must have a known Gleason sum based on biopsy or TURP at the time of registration.
3. Locally Resectable Disease: Patients must have disease (localized or locally advanced) which is deemed by the surgeon to be resectable. Lymph node metastasis or lymph nodes suspicious of harboring metastasis should be deemed surgically resectable by the surgeon.
4. Determination of high-risk status: Patients must have either: 1) a Prostate biopsy Gleason sum >/= 8 OR 2) PSA >/= 20.
5. Prior Treatment: No prior treatment for prostate cancer including prior surgery (excluding TURP), pelvic lymph node dissection, radiation therapy, or chemotherapy. Patients who have initiated leuprolide acetate within 1 week of signing consent will be eligible.
6. Patients must be appropriate candidates for radical prostatectomy. Evidence of underlying cardiac disease should be evaluated prior to enrollment to ensure that patients are not at high risk of cardiac complications.
7. ECOG performance status of 0 or 1;
8. Required values for initial laboratory tests: a) WBC >/= 3000/uL; b) ANC >/= 1500/uL, c) Platelets >/= 100 x 10^3/uL; d) Hemoglobin >/= 9 g/dL; e) Creatinine </= 2.0 x ULN; f) AST </= 2.5 x ULN; g) Bilirubin 0 - 1.0 mg/dL, except patients with Gilbert's Syndrome, who must have a total bilirubin less than 3.0 mg/mL;
9. Men >/= 18 years of age
10. Patients must agree to practice barrier birth control methods while on therapy, prior to surgery.

Exclusion Criteria:

1. Any other malignancy from which the patient has been disease-free for less than 5 years, with the exception of adequately treated and cured basal or squamous cell skin cancer.
2. Autoimmune disease: Patients with a history of Inflammatory Bowel Disease (including Crohn's disease and ulcerative colitis) are excluded from this study as are patients with a history of autoimmune disease (e.g., rheumatoid arthritis, systemic progressive sclerosis [scleroderma], Systemic Lupus Erythematosus, autoimmune vasculitis [e.g., Wegener's Granulomatosis]).
3. Known HIV or chronic hepatitis.
4. Any underlying medical condition, which in the opinion of the Investigator, will make the administration of study drug hazardous or obscure the interpretation of adverse events, such as a condition associated with frequent diarrhea.
5. Patients who have had a history of acute diverticulitis, intra-abdominal abscess, GI obstruction, abdominal carcinomatosis which are known risks factors for bowel perforation, should be excluded from the study.
6. Any non-oncology vaccine therapy used for prevention of infectious diseases (for up to one month prior to or after any dose of ipilimumab.
7. Concomitant therapy with any of the following: IL-2, interferon or other non-study immunotherapy regimens; cytotoxic chemotherapy; immunosuppressive agents; other investigation therapies; or chronic use of systemic corticosteroids (used in the management of cancer or non-cancer-related illnesses);
8. Previous treatment with other investigational products within 30 days;
9. Previous enrollment in another MDX-010 (BMS-734016) clinical trial or prior treatment with a CD137 agonist or CTLA-4 inhibitor or agonist
10. Concurrent use of 5-alpha-reductase inhibitors (finasteride, dutasteride).
11. Prisoners or patients who are compulsorily detained (involuntarily incarcerated) for treatment of either a psychiatric or physical (e.g., infectious disease) illness must not be enrolled in this study.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2010-09; Primary Completion 2015-10 (Actual); Study Completion 2015-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Padmanee Sharma, MD, PHD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- University of Texas MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment period: September 1, 2010 to June 5, 2013. All recruitment done at The University of Texas MD Anderson Cancer Center.
Period: Overall Study
Arm/Group | Neoadjuvant Ipilimumab
Started | 19
Completed | 16
Not Completed | 3
Not completed — Withdrawal by Subject | 1
Not completed — Ineligible, Screen Failure | 1
Not completed — Death | 1

BASELINE CHARACTERISTICS:
Population: Two participants are not included in the demographics, excluded from the study due to screening failure or withdraw prior to being assigned any treatment.
Arm/Group | Neoadjuvant Ipilimumab
Number analyzed (Participants) | 17
Age, Continuous [Mean (Full Range); unit: years] | 57.9 [36 to 71]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 17
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 14
  Black | 3
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 17
PSA (Average) Tumor Clinical Stage [Count of Participants; unit: Participants] — Prostate-specific antigen (PSA) 4 categories for describing the local extent of a prostate tumor, ranging from T1 to T4
  Participants
    T1 | 5
    T2 | 4
    T3 | 8
Gleason Score [Count of Participants; unit: Participants]
  7 | 1
  8 | 5
  9 | 10
  10 | 1
Lupron Ipilimumab Dose [Count of Participants; unit: Participants]
  One dose | 1
  Two doses | 16
Surgery [Count of Participants; unit: Participants]
  Yes | 16
  No | 1

OUTCOME MEASURES:

1. Primary Outcome: Immunologic Response: Number of Participants With Immune Response
Description: Immunological response assays were measured at several time points starting at baseline until the eighth week after starting the medicine for each participant. The immunological responses measured were Cluster of Differentiation 4 (CD4), Cluster of Differentiation 8 (CD8) and Inducible T-cell Costimulatory (ICOS) markers. T-cells with the CD4 marker help coordinate the immune system response to an invader. Killer T-cells have the CD8 marker and are responsible for killing the invader. ICOS is a molecule which stimulates the activity of the immune response of the killer T-Cells and memory T cells. Participants with at least a 2 fold increase in the presence of CD4, CD8, or ICOS markers from the participant's baseline measure were considered a responder for that marker.
Time Frame: Baseline to Week 8
Population: One participant was not evaluable for outcome due to early death. Of evaluable 16 participants, the number of participants (N) analyzed reflected in CD4, CD8 and ICOS that are associated with immune response.
Measure: Count of Participants; unit: Participants
Arm/Group | Neoadjuvant Ipilimumab
Number analyzed (Participants) | 16
Participants
  CD4: number analyzed (Participants) | 15
  CD4 | 12
  CD8: number analyzed (Participants) | 14
  CD8 | 7
  ICOS: number analyzed (Participants) | 14
  ICOS | 9

ADVERSE EVENTS:
Time Frame: Adverse event collection from baseline until 30 days after the last dose of drug, approximately 14 weeks post surgery.
Description: Two participants of nineteen registered on the study were excluded prior to any treatment assignment due to screen failure and withdrawal, therefore are not included in adverse event reporting.
Arm/Group | Neoadjuvant Ipilimumab
All-Cause Mortality (participants affected / at risk) | 1/17
Serious Adverse Events (participants affected / at risk) | 2/17
Other Adverse Events (participants affected / at risk) | 17/17
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Neoadjuvant Ipilimumab (N=17)
Bilateral pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Cardiac arrest (Cardiac disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Neoadjuvant Ipilimumab (N=17)
Cardiac arrest (Cardiac disorders) | 1
Acute respiratory distress syndrome (ARDS) (Respiratory, thoracic and mediastinal disorders) | 1
Rash (Skin and subcutaneous tissue disorders) | 9
Fatigue (General disorders) | 8
Transaminitis (Investigations) | 7
Colitis/Diarrhea (Gastrointestinal disorders) | 9
Headache (General disorders) | 6
Pancreatitis (Gastrointestinal disorders) | 5
Hypophysitis (Investigations) | 5
Fever (General disorders) | 1
Dehydration (Metabolism and nutrition disorders) | 2
Synocope (Nervous system disorders) | 1
Hypoalbuminemia (Metabolism and nutrition disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes